CLINICAL TRIAL: NCT02708277
Title: Reproductive Outcome Affected by Two Adjunctive Treatments in Patients With Infertility Due to Severe Intrauterine Adhesions.
Brief Title: Reproductive Outcome Affected by Two Adjunctive Treatments in Patients With Severe Intrauterine Adhesions
Acronym: ROABTIPWSIUA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuqing Chen (Other)
Responsible Party: Sponsor-Investigator, Yuqing Chen, Associate chief physician, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUA-21
Record Dates: First submitted 2016-03-04; First posted 2016-03-15 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Asherman's Syndrome
Keywords: intrauterine contraceptive device; intrauterine balloon
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): At the end of the procedure the surgery loop-shaped intrauterine contraceptive device (IUCD) was placed in the uterine cavity.
  Interventions: Device: loop-shaped intrauterine contraceptive device
- Group B (Experimental): At the end of the procedure the surgery an intrauterine balloon (Cook Medical) was placed in the uterine cavity.
  Interventions: Device: intrauterine balloon (Cook Medical)

INTERVENTIONS:
Device: loop-shaped intrauterine contraceptive device — Intrauterine contraceptive device can temporary protective layer between the endometrium wound during the most critical three weeks after the surgery to prevent adhesion reformation.
  Arms: Group A
Device: intrauterine balloon (Cook Medical) — The balloons used in this study is heart- shaped that resembled the shape of the uterine cavity and could fully separate the two sides of the uterine wall and the corners of the uterus compare to loop-shaped intrauterine contraceptive device.
  Arms: Group B

SUMMARY:
The purpose of this study is to compare the outcome of loop intrauterine contraceptive device and heart-shaped intrauterine balloon for the adjunctive treatment of severe intrauterine adhesions in patients with infertility.

DETAILED DESCRIPTION:
Intrauterine adhesion, also known as Asherman's syndrome, is the partial or complete occlusion of the uterine cavity as a result of endometrium damage. Most intrauterine adhesions patients manifest amenorrhea, reduced menstrual pattern, infertility, and intrauterine growth restriction, which seriously affect their reproductive health. Currently, hysteroscopy is the preferred method of intrauterine adhesions diagnosis and treatment. However, because intrauterine adhesions patients generally have poor endometrium repair capability, the incidence rate of reformation of intrauterine adhesions ranging from 20%-62.5% in those with severe adhesions. The successful pregnancy rate after treatment in severe Asherman's syndrome is reported to be consistently lower, only 33%. The prevention of intrauterine adhesions recurrence after trans-cervical resection of adhesion is clinically important but difficult. Therefore, this study was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe intrauterine adhesions
* infertility

Exclusion Criteria:

* endometrial tuberculosis
* grossly abnormal semen analysis
* ovarian failure, hydrosalpinx fluid
* patients who did not proceed to second-look hysteroscopy within the specified time frame
* Women with no desire to pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuzhong Yao, professor, Study Director — First Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Orhue AA, Aziken ME, Igbefoh JO. A comparison of two adjunctive treatments for intrauterine adhesions following lysis. Int J Gynaecol Obstet. 2003 Jul;82(1):49-56. doi: 10.1016/s0020-7292(03)00030-4. PMID 12834941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2011 to February 2013, women with severe intrauterine adhesions who presented with a history of infertility were initially included in the study.
Pre-assignment Details: Exclusion criteria: endometrial tuberculosis, grossly abnormal semen analysis, ovarian failure, hydrosalpinx fluid, and patients who did not proceed to second-look hysteroscopy within the specified time frame，women with no desire to pregnancy.
Groups:
- Loop-shaped Intrauterine Device Group: At the end of the procedure the surgery loop-shaped intrauterine contraceptive device (IUCD) was placed in the uterine cavity.
  loop-shaped intrauterine contraceptive device: Intrauterine contraceptive device can temporary protective layer between the endometrium wound during the most critical three weeks after the surgery to prevent adhesion reformation.
- Intrauterine Balloon Group: At the end of the procedure the surgery an intrauterine balloon (Cook Medical) was placed in the uterine cavity.
  intrauterine balloon (Cook Medical): The balloons used in this study is heart- shaped that resembled the shape of the uterine cavity and could fully separate the two sides of the uterine wall and the corners of the uterus compare to loop-shaped intrauterine contraceptive device.
Period: Overall Study
Arm/Group | Loop-shaped Intrauterine Device Group | Intrauterine Balloon Group
Started | 50 | 43
Completed | 43 | 39
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 43 | 39 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 39 | 82
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (4.3) | 31.6 (4.3) | 31.9 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 43 | 39 | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pregnancy in Loop-shaped Intrauterine Device Group and Intrauterine Balloon Group
Time Frame: three years
Measure: Number; unit: participants
Arm/Group | Loop-shaped Intrauterine Device Group | Intrauterine Balloon Group
Number analyzed (Participants) | 43 | 39
participants | 12 | 22
Statistical Analysis 1: Comparison: Loop-shaped Intrauterine Device Group vs Intrauterine Balloon Group; Test type: Superiority or Other; p = 0.009, Chi-squared

2. Secondary Outcome: Menstruation Pattern(Improvement or No Significant Change) of All Participants
Description: Comparing with preoperative and postoperative menstrual duration, numbers of sanitary napkin using and wet area ratio of sanitary napkin to judgment whether menstrual quantity is improvement in patients
Time Frame: Within the first 3 months after surgery
Measure: Number; unit: participants
Arm/Group | Loop-shaped Intrauterine Device Group | Intrauterine Balloon Group
Number analyzed (Participants) | 43 | 39
participants
  Menstruation pattern improvement | 35 | 28
  Menstruation pattern no significant change | 8 | 11
Statistical Analysis 1: Comparison: Loop-shaped Intrauterine Device Group vs Intrauterine Balloon Group; Test type: Superiority or Other; p = 0.303, Chi-squared

3. Secondary Outcome: Endometrial Thickness of All Participants in the Mid Menstrual Measured by Color Doppler Ultrasound
Time Frame: Within the first 3 months after surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Loop-shaped Intrauterine Device Group | Intrauterine Balloon Group
Number analyzed (Participants) | 43 | 39
mm | 6.1 (1.8) | 6.1 (1.7)
Statistical Analysis 1: Comparison: Loop-shaped Intrauterine Device Group vs Intrauterine Balloon Group; Test type: Superiority or Other; p = 0.606, t-test, 2 sided

4. Secondary Outcome: Number of Participants With Reformation of Intrauterine Adhesions in Loop-shaped Intrauterine Device Group and Intrauterine Balloon Group
Time Frame: Within the first 3 months after surgery
Measure: Number; unit: participants
Arm/Group | Loop-shaped Intrauterine Device Group | Intrauterine Balloon Group
Number analyzed (Participants) | 43 | 39
participants
  Reformation of intrauterine adhesions | 16 | 6
  Peripheral adhesions | 13 | 4
  Central adhesions | 1 | 2
  Mixed adhesions | 2 | 0
Statistical Analysis 1: Comparison: Loop-shaped Intrauterine Device Group vs Intrauterine Balloon Group; Test type: Superiority or Other; p = 0.05, Chi-squared

ADVERSE EVENTS:
Arm/Group | Loop-shaped Intrauterine Device Group | Intrauterine Balloon Group
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/39
Other Adverse Events (participants affected / at risk) | 1/43 | 1/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loop-shaped Intrauterine Device Group (N=43) | Intrauterine Balloon Group (N=39)
vaginitis (Infections and infestations) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was conducted in a university hospital.If this was a multicenter study, the results should be more reasonable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No